CLINICAL TRIAL: NCT06169059
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Multiple Administration of JC-013 and JLP-2004 in Healthy Adult Volunteers
Brief Title: To Evaluate the Safety and Pharmacokinetic Characteristics After Multiple Administration of JC-013 and JLP-2004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP-2004-101
Record Dates: First submitted 2023-11-20; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment(Experimental): JLP-2004 (Experimental): Group I(Peroid I-comparator, Peroid II-JLP-2004), Group II(Period I-JLP-2004, Period II-Comparator)
  Interventions: Drug: JLP-2004; Drug: JC-013
- Control(Active Comparator): JC-013 (Active Comparator): Group I(Peroid I-comparator, Peroid II-JLP-2004), Group II(Period I-JLP-2004, Period II-Comparator)
  Interventions: Drug: JLP-2004; Drug: JC-013

INTERVENTIONS:
Drug: JLP-2004 — administration of JLP-2004(COX-2 inhibitor)
Drug: JC-013 — administration of JC-013(COX-2 inhibitor))

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics after multiple administration of JC-013 and JLP-2004

DETAILED DESCRIPTION:
A phase 1 clinical trial to compare and evaluate the safety and pharmacokinetic characteristics after multiple administration of JC-013 and JLP-2004 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 years or older at the time of screening
2. At the time of screening, those who weigh more than 50.0 kg and have a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.
3. Those who do not have congenital or chronic diseases and have no pathological symptoms or findings as a result of internal medical examination (if necessary, electroencephalography, electrocardiogram, chest and stomach endoscopy, or gastrointestinal radiography)
4. Those who be considered suitable for clinical subjects according to the results of laboratory tests (hematology tests, blood chemistry tests, urine tests, serum tests, blood coagulation tests, urine drugs tests), physical examinations and 12-lead electrocardiography at the time of screening
5. Those who voluntarily decide to participate and agree in writing to comply with the subject compliance requirements during the clinical trial period after receiving a detailed explanation of this clinical trial and fully understanding it

Exclusion Criteria:

1. Those who have current or past medical history of clinically significant liver, kidney, nervous system, mental, respiratory, endocrine, blood disease, tumor, genitourinary, cardiovascular, digestive, and musculoskeletal systems, as well as the following symptoms or history.

   ① Renal impairment

   ② Liver disorder
2. For women, pregnant women (Urine-HCG positive) or breastfeeding mother
3. Those who have clinically significant hypersensitivity reactions such as asthma, hives, allergies, etc. to the main ingredient (Pelubiprofen), additives, or other drugs (aspirin or other non-steroidal anti-inflammatory drugs (including COX-2 inhibitors)) and have a history of hypersensitivity reaction
4. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
5. Those with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of clinical trial drugs

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
AUC last of JLP-2004 | 24 hours
Cmax of JLP-2004 | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea